CLINICAL TRIAL: NCT06300541
Title: Prevalence and Impact of Sarcopenia in Patients With Inflammatory Bowel Disease and the Significance of Removing the Colon
Brief Title: Prevalence and Impact of Sarcopenia in Patients With Inflammatory Bowel Disease
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Ersta Hospital, Sweden (Other)
Responsible Party: Principal Investigator, Jonas Varkey, Principal investigator, Senior Consultant, MD, PhD,, Sahlgrenska University Hospital
Other Study IDs: 940730
Record Dates: First submitted 2024-02-01; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Inflammatory Bowel Diseases; Sarcopenia
Keywords: sarcopenia
MeSH Terms: conditions — Inflammatory Bowel Diseases; Sarcopenia | interventions — Colectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, feces, tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1) IBD conventional treatment,: Medical therapy
  Interventions: Procedure: Colectomy
- 2) Colectomy: Surgical treatment
  Interventions: Procedure: Colectomy

INTERVENTIONS:
Procedure: Colectomy — Observational study.

SUMMARY:
Sarcopenia is a condition characterized by significant muscle loss resulting in impaired muscle function. This condition is likely associated with a biological deviation leading to reduced reserves to withstand stressors, resulting in a poorer prognosis. The incidence of sarcopenia among patients with inflammatory bowel diseases (Ulcerative Colitis and Crohn's disease) is currently approximately 40-60%. This is likely a consequence of the preference for drug treatment over surgery, while many patients have continuous inflammation in their intestines leading to muscle loss and subsequently increased morbidity and mortality.

The purpose of the study is to identify the prevalence of sarcopenia among patients experiencing a severe flare-up of their bowel disease and to evaluate whether the removal of the colon results in improved nutritional status. Furthermore, the investigators aim to investigate whether there is a specific microbiota composition related to an unfavorable course.

The participants are longitudinally monitored with measurements taken at the flare-up/before surgery and one year afterward, including body composition, function, dietary recording, quality of life, blood tests, fecal samples, and intestinal biopsies that will be analyzed. The investigators plan to correlate body composition with a biological profile and then evaluate if there is an association. Additionally, the investigators aim to analyze if these markers are linked to different outcomes after colectomy. This study will contribute to an enhanced understanding of patients with advanced IBD and possibly change the perspective on how the clinicians should prioritize these patients for surgery. The investigators believe this study will lead to an improvement in healthcare quality and an enhanced understanding of how these disease processes function.

DETAILED DESCRIPTION:
All examinations and laboratory tests will be conducted on two occasions. Moreover, two cohorts will be present. That is, one group where participants experiencing a severe flare-up receive medical treatment, and another group where participants with the bowel disease undergo surgery. All samples/examinations and surveys are therefore done before the operation/during the flare-up, and then again one year later during a follow-up assessment

ELIGIBILITY:
Inclusion Criteria:

* All adult patients experiencing an acute flare-up of their bowel disease (ulcerative colitis or Crohn's disease) admitted to a hospital in the Region Västra Götaland and Stockholm are invited to participate in the study.

Exclusion Criteria:

* Not wishing to participate in the study Inability to understand the language or study procedures

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with severe IBD.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with increase in muscle mass as assessed by DEXA scan. | 1 year
  The primary outcome measure is to compare the changes in muscle mass, as quantified by DEXA, between baseline and the 1-year follow-up in participants who have undergone either colectomy or medical treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Varkey, MD. Ph D, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No